CLINICAL TRIAL: NCT03642418
Title: User-Friendly Spirometer and Mobile App for Self-Management and Home Monitoring of Asthma Patients Phase 2
Brief Title: User-Friendly Spirometer and Mobile App for Self-Management and Home Monitoring of Asthma Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 17-22946
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Asthma Acute; Asthma in Children; Asthma Chronic; Asthma Attack
Keywords: asthma, children, spirometry, lung function, asthma action plan, asthma exacerbation, self management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this proposal is to use an in-home, smartphone-enabled, hand-held spirometer to determine the FEV1% predicted ranges that predict the Yellow Zone threshold.

DETAILED DESCRIPTION:
The study hypothesizes that objective lung function tracking at-home, using a portable spirometer in addition to conventional symptom monitoring (in which asthmatic patients self-report and track their own symptoms), will result in more reliable detection of exacerbation in children 6-15 years old with asthma.

This is a 44-week, single arm, blinded nonrandomized trial to determine clinically relevant ranges in FEV1% predicted that correlate with the Yellow Zone of the Asthma Action Plan.

A total of 100 pediatric subjects (between the ages of 6 and 15 years old) with physician-diagnosed mild or moderate persistent asthma treated on controller therapy will be enrolled from the ED, Inpatient Units, Pulmonary Medicine Clinic, and Allergy/Immunology Clinic at UCSF Benioff Children's Hospital San Francisco.

Primary Specific Aim

To determine the FEV1% predicted changes that correspond with a change from the Green to Yellow Zone.

The primary outcome will be Yellow Zone episodes, as identified by the occurence of any of the following:

Symptom Diary score > 4 ATAQ score > 1

Secondary Specific Aim

To determine the FEV1% predicted changes that correspond with a change from the Yellow to Red Zone.

The secondary outcome will Red Zone episodes, as identified by the occurence of any of the following:

ED or Urgent Care visit Administration of systemic (oral, IM, or IV) corticosteroids Hospitalization

ELIGIBILITY:
Inclusion Criteria:

1. Physician-diagnosed mild or moderate persistent asthma
2. On controller therapy [inhaled corticosteroid (ICS), ICS + leukotriene receptor antagonist (LTRA), or ICS + long-acting beta agonist (LABA)] for at least the previous six months
3. At least one severe exacerbation requiring systemic corticosteroids in the previous year
4. Baseline FEV1 >/= 70% predicted for age, gender, and height according to published reference standards
5. Parental consent and the child's assent

Exclusion Criteria:

1. Chronic obstructive respiratory disorder other than asthma (e.g., cystic fibrosis, primary ciliary dyskinesia)
2. Severe persistent asthma, as evidenced by any of the following:

   * 3 hospitalizations
   * 6 severe exacerbations in the previous year on chronic oral corticosteroid therapy daily symptoms
3. Inability to perform acceptable spirometry
4. History of collapsed lung
5. History of syncope with forced exhalation
6. Not owning an iOS™ device (e.g., iPhone®, iPod®, or iPad®)
7. Lacking access to wireless local area networking (Wi-Fi™)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 6 to15 years old with mild to moderate persistent asthma seen in the outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Yellow Zone episodes | 44 weeks
  defined by the occurrence of any of the following: (1) Symptom Diary score > 4 and (2) ATAQ score > 1

SECONDARY OUTCOMES:
Red Zone episodes | 44 weeks
  defined by the occurrence of any of the following:
  ED or Urgent Care visit Administration of systemic (oral, IM, or IV) corticosteroids Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ngoc P Ly, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF- Benioff Children Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No